CLINICAL TRIAL: NCT07001774
Title: Vitalis Cardio Pilot Study: A Single Arm Efficacy Study of a Clinical Health Coaching Model
Brief Title: Vitalis Cardio Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lucas Carr (Other)
Collaborators: Google LLC. (Industry)
Responsible Party: Sponsor-Investigator, Lucas Carr, Associate Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 202308018
Record Dates: First submitted 2024-12-19; First posted 2025-06-03 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2024-11

CONDITIONS: Cardiovascular Disease Risk Factor
Keywords: health coaching; cardiovascular disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vitalis Cardio Intervention (Experimental): The intervention includes health coaching, health education, and wearable activity monitoring.
  Interventions: Behavioral: Vitalis Cardio

INTERVENTIONS:
Behavioral: Vitalis Cardio — Participants receive five free health coaching sessions with a trained student health coach, access to two health education videos, and a free wrist worn activity monitor to keep track of their physical activity and sleep behaviors.

SUMMARY:
The objective of this study was to evaluate the efficacy and feasibility of a 12-week behavioral counseling intervention that has been integrated into the primary care setting on psychosocial, behavioral, and health outcomes in a large sample of adults with at least one CVD risk factor.

Aim 1: Evaluate the efficacy of a 12-week behavioral counseling intervention on psychosocial outcomes of adults with at least one CVD risk factor.

H1: We hypothesize participants will improve their behavioral regulation skills and habit formation skills over 12 weeks.

Aim 2: Evaluate the efficacy of a 12-week behavioral counseling intervention on behavioral outcomes (physical activity, diet, and sleep) of adults with at least one CVD risk factor.

H2: We hypothesize participants will improve PA (daily steps), diet (total daily kilocalories), and sleep (sleep time, sleep efficiency) over the 12-week intervention.

Aim 3: Evaluate the efficacy of a 12-week behavioral counseling intervention on health outcomes (blood pressure, weight, waist circumference, body composition, quality of life) of adults with at least one CVD risk factor.

H3: We hypothesize participants will improve blood pressure, weight, waist circumference, body composition, quality of life over the 12-week intervention.

DETAILED DESCRIPTION:
The U.S. Preventive Services Task Force (USPSTF) issued a Grade B level recommendation (moderate net benefit) that healthcare providers offer PA and dietary behavioral counseling interventions to adults with known CVD risk factors. Unfortunately, these types of programs are rarely implemented in the healthcare setting. Consistent with the USPSTF recommendations, the American College of Sports Medicine's Exercise is Medicine (EIM) initiative has called for PA to be integrated into healthcare by screening all patients for inactivity and providing inactive patients with behavioral counseling resources. Our team has established an evidence-based EIM program that screens patients for inactivity and connects them to a behavioral counseling program. In November 2018, Family Medicine well-visit patients started receiving screening for inactivity using the two-item Exercise Vital Sign (EVS) questionnaire. In 2021, the first Health Coaching training program was developed in the state of Iowa that is recognized by the National Board for Health and Wellness Coaching (NBHWC). In June 2023, a new clinical workflow was launched in the university electronic medical record system (Epic) which streamlines the process of connecting inactive Family Medicine patients with local health coaches.

This study will test the efficacy of a behavioral counseling program on targeted health behaviors and cardiometabolic risk factors among a sample of adults who are at increased risk for cardiovascular disease.

Patients being treated in the Family Medicine clinic who report wanting to meet with a health coach will be provided a link to an online Health Coach Request form in their After Visit Summary report and MyChart accounts. Patients who choose to open and complete the online Health Coach Request form provide their contact information in the form. Interested patients will be contacted via email to gauge their interest and eligibility. Eligible patients will be enrolled into a 12 week intervention that includes meeting with a student health coach 5 times over 12 weeks, wearing an activity monitor daily, and watching two health education videos.

Aim 1: Evaluate the efficacy of a 12-week behavioral counseling intervention on psychosocial outcomes of adults with at least one CVD risk factor.

Aim 2: Evaluate the efficacy of a 12-week behavioral counseling intervention on behavioral outcomes (physical activity, diet, and sleep) of adults with at least one CVD risk factor.

Aim 3: Evaluate the efficacy of a 12-week behavioral counseling intervention on health outcomes (blood pressure, weight, waist circumference, body composition, quality of life) of adults with at least one CVD risk factor.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults between 18 and 80 years old

  * Report at least one known cardiovascular disease risk factor (high blood pressure (systolic > 130 or diastolic > 80), high low-density lipoprotein cholesterol (>160), diabetes diagnosis, smoking, obesity (BMI>30.0), or physical inactivity (<150 minutes/week of moderate intensity physical activity)
  * Physically able to become more active
  * Own a smartphone with a data plan
  * Able to understand English and provide informed consent Report intentions to improve either physical activity, eating, or sleep behaviors Requesting a health coach

Exclusion Criteria:

* • Unable to become more active

  * Does not own a smartphone with a data plan
  * Inability to read, complete or sign the consent form and survey
  * Presence of a psychiatric disorder that is not managed/unstable or suicidal ideation/actuation in preceding 12 months Pregnant or plan to become pregnant in the next 2 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-09-19 (Actual); Primary Completion 2025-08-11 (Actual); Study Completion 2025-08-11 (Actual)

PRIMARY OUTCOMES:
Behavioral Regulation Skills | From enrollment to 12 weeks
  Participant's perceived ability to regulate their physical activity, diet, and sleep behaviors using a six item survey that uses a 5 point Likert scale. Scores will range from 6 (low skills) to 30 (high skills).
Habit formation skills | From enrollment to 12 weeks
  Habit formation will be measured with a 3 question survey using a 5 point likert scale. Responses will range from 3 (weak habit) to 15 (strong habit).

SECONDARY OUTCOMES:
Physical activity | From enrollment to 12 weeks
  Daily steps will be measured for 7 days with a Fitbit activity monitor
Diet behavior | From enrollment to 12 weeks
  Measured with the Automated Self-Administered Dietary Assessment (ASA2$) Tool
Sleep behavior | From enrollment to 12 weeks
  Sleep time and sleep efficiency will be measured for 7 days with a Fitbit activity monitor
Global Health | From enrollment to 12 weeks
  Measured with two questions on a 5 point likert scale. Scores will range from 2 (poor) to 10 (excellent)
Weight (lbs) | From enrollment to 12 weeks
  Weight will be measured to the nearest 0.5 lb with a medical scale

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No